CLINICAL TRIAL: NCT06294899
Title: Evaluation of Point-of-Care Ultrasound Along With C-Reactive Protein-Point of Care Tests Impact on Clinical Decision-making and Perceived Usefulness in Routine Healthcare Use in Patients With Lower Respiratory Tract Infection. Correlation Between C-Reactive Protein Concentrations and Lung Ultrasound Findings.
Brief Title: CRP and Lung Ultrasound in Respiratory Evaluation
Acronym: PLURE
Status: Not yet recruiting | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Anna Llinas Vaquer, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: 23/222-P
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Primary Health Care; Lower Respiratory Tract Infection
Keywords: C-Reactive Protein; Lung ultrasonography; Lower Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound will be performed to patients with suspected lower respiratory tract infections.
Diagnostic Test: C-Reactive Protein Test — C-Reactive Protein Test will be performed to patients with suspected lower respiratory tract infections.

SUMMARY:
Lower respiratory tract infections (LRTIs) are one of the most common reasons for consultation in Primary Care centres. Differentiating between viral and bacterial aetiologies can be challenging, leading to inappropriate antibiotic prescribing. Lung ultrasound (LUS), an imaging test that gained particular relevance since the beginning of the SARS-CoV-2 pandemic, offers several advantages over the classic chest X-ray in detecting and monitoring LRTIs, especially when pleural involvement exists.

This study aims to correlate LUS findings with capillary blood C-Reactive Protein (CRP) values in patients with LRTIs, evaluating LUS as a diagnostic tool and its impact on therapeutic decisions. The descriptive observational study, conducted from January 2024 to December 2026 in Lleida, will include LRTI patients attending Primary Care centres. By validating LUS as a rapid and non-invasive diagnostic tool, unnecessary antibiotic prescriptions can be reduced, promoting LUS as a complementary test in Primary Care consultations. This will facilitate appropriate diagnosis and treatment decisions for patients with LRTIs, enhancing the overall management of respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Clinical suspicion of LRTI defined as acute illness lasting less than 21 days, with cough as the main symptom, accompanied by at least one other lower respiratory symptom (such as sputum production, dyspnoea, difficult breathing, or chest pain) without any other explanation for the clinical picture.
* Ability to read, understand and willingness to give written consent to participate in the study.

Exclusion Criteria:

* Patients who have been treated with antibiotics during the last 14 days up to inclusion.
* Patients with hemodynamic instability or that need emergency medical care due to the current clinical condition.
* Previous diagnosis of lung or pleural cancer.
* Thoracic surgery within the past 60 days.
* Lung interstitial diseases.
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower respiratory tract infections attending Primary Care centres in Lleida.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound patterns | Each evaluation will be carried out during a dedicated ultrasound session, with an approximate duration of 15 minutes per participant.
  Standardized criteria will be used to differentiate between normal patterns and those that may indicate pathological conditions. The classification of patterns will include, but not be limited to, tissue heterogeneity, presence of masses or fluids, and characteristics of the edges of lesions.
C-Reactive Protein | CRP levels will be measured at baseline.
  This metric assesses the levels of C-Reactive Protein in the blood, an indicator of inflammation in lower respiratory tract infections already used in the Primary Care practice.

IPD SHARING:
Plan to Share IPD: No